CLINICAL TRIAL: NCT03294681
Title: Trans-impedance Matrix
Brief Title: Collection and Characterization of Objective Measures to Explore the Specificity of Algorithms
Status: Completed | Type: Observational
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Other Study IDs: CLTD5676
Record Dates: First submitted 2017-09-15; First posted 2017-09-27 (Actual); Results first posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cochlear Implant Recipients
  Interventions: Device: Objective measures with CSEP

INTERVENTIONS:
Device: Objective measures with CSEP — Objective measures to be conducted with Custom SoundTM EP 5 software and the CP900 series sound processor in CI532 and CI512 Cochlear Implant recipients

SUMMARY:
The aim of this descriptive study is to collect and describe the characteristics of objective measures to explore the specificity of algorithms.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for cochlear implantation with the CI532 or CI512 devices
* 18 years of age or older at the time of enrolment
* Normal cochlea anatomy, established via pre-operative Computer Tomography
* Willingness to participate in and to comply with all requirements of the protocol

Exclusion Criteria:

* Prior cochlear implantation in the ear to be implanted
* Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array
* Abnormal cochlear anatomy on pre-operative Computer Tomography or Magnetic Resonance Imaging
* Additional handicaps that would prevent participation in evaluations
* Pregnant and breast feeding women, prisoners, or anyone in custody
* Unrealistic expectations on the part of the subject, regarding the possible benefits, risks and limitations that are inherent to the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Routine patients undergoing a standard cochlear implantation.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Volckaerts, PhD, Study Director — Cochlear
Locations (6):
- HEARing CRC, Carlton, Australia
- Germany (3):
  - Hals-Nasen-Ohren-Klinik Universitätsklinikum Erlangen, Erlangen
  - Klinik für Hals-, Nasen-, Ohrenheilkunde Universitätsklinikum Frankfurt Goethe-Universität, Frankfurt am Main
  - Universitätsklinikum Schleswig- Holstein - Campus Kiel Klinik für Hals-, Nasen-, Ohrenheilkunde, Kopf- und Halschirurgie, Kiel
- Spain (2):
  - Complejo Hospitalario Universitario Insular Materno Infantil, Las Palmas de Gran Canaria
  - Clinica Universitaria de Navarra, Pamplona

REFERENCES:
- [Derived] Hoppe U, Brademann G, Stover T, Ramos de Miguel A, Cowan R, Manrique M, Falcon-Gonzalez JC, Hey M, Baumann U, Huarte A, Liebscher T, Bennett C, English R, Neben N, Ramos Macias A. Evaluation of a Transimpedance Matrix Algorithm to Detect Anomalous Cochlear Implant Electrode Position. Audiol Neurootol. 2022;27(5):347-355. doi: 10.1159/000523784. Epub 2022 Mar 18. PMID 35306487

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 153 participants were recruited in six centres from 03 October 2017 to 29 May 2019.
Groups:
- Cochlear Implant Recipients: CI532 and CI512 cochlear implant recipients
Period: Overall Study
Arm/Group | Cochlear Implant Recipients
Started | 153
Completed | 152
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 153 participants were recruited and one patient withdrew consent. The data of this participant were not analyzed.
Arm/Group | Cochlear Implant Recipients
Number analyzed (Participants) | 152
Age, Continuous [Mean (Full Range); unit: years] | 58 [19 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 73
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 9
  Germany | 115
  Spain | 28

OUTCOME MEASURES:

1. Primary Outcome: Specificity (%) of Transimpedance Measurement to Identify Electrode Fold-over
Description: Measured with Custom SoundTM EP 5. It took one minute to measure all electrodes in surgery.
  Intraoperative transimpedance measures from 148 ears without fold-overs (as evidenced by radiographic imaging) were analysed to assess the specificity of the algorithm.
Time Frame: at surgery, within one minute
Population: 148 ears were analyzed from 145 participants (with three bilateral participants providing 148 ears). From the 152 baseline participants, seven were excluded from the analysis: for three participants, no transimpedance data were obtained intra-operatively and for four participants the transimpedance data showed measurement abnormalities.
Measure: Number (90% Confidence Interval); unit: Percentage of ears
Units Other Than Participants: ears
Arm/Group | Cochlear Implant Recipients
Number analyzed (Participants) | 145
Number analyzed (ears) | 148
Percentage of ears | 98.6 [95.8 to 99.75]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Cochlear Implant Recipients
All-Cause Mortality (participants affected / at risk) | 0/153
Serious Adverse Events (participants affected / at risk) | 2/153
Other Adverse Events (participants affected / at risk) | 0/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cochlear Implant Recipients (N=153)
Renal carcinoma (Renal and urinary disorders) | 1 (1)
Pass out related to heat (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators can publish and/or present their own data and process their data with their own algorithms. At study end 2 joint publications by the clinical investigators/sponsor are planned with the Coordinating Investigator writing the publication. All abstract/publication must be reviewed by the sponsor at least 30 days in advance. If a publication contains information that the sponsor finds worth protecting the sponsor has the right to delay the publication/presentation for 90 days.

DOCUMENTS (2):
  • Study Protocol (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/81/NCT03294681/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/81/NCT03294681/SAP_001.pdf